CLINICAL TRIAL: NCT03164135
Title: Safety and Feasibility Study of Allotransplantation of CRISPR/Cas9 CCR5 Gene Modified CD34+ Hematopoietic Stem/Progenitor Cells in HIV-infected Subjects With Hematological Malignances
Brief Title: Safety of Transplantation of CRISPR CCR5 Modified CD34+ Cells in HIV-infected Subjects With Hematological Malignances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Peking University (Other); Capital Medical University (Other)
Responsible Party: Principal Investigator, Chen Hu, Study Director, Affiliated Hospital to Academy of Military Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-HSPC-R5
Record Dates: First submitted 2017-05-18; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Intervention Model Description: CD34+ hematopoietic stem/progenitor cells from donor are treated with CRISPR/Cas9 before transplantation into the patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCR5 gene modification (Experimental): CD34+ hematopoietic stem/progenitor cells from donor are treated with CRISPR/Cas9 before transplantation into the patient.
  Interventions: Genetic: CCR5 gene modification

INTERVENTIONS:
Genetic: CCR5 gene modification — CD34+ hematopoietic stem/progenitor cells from donor are treated with CRISPR/Cas9 targeting CCR5 gene.

SUMMARY:
The investigators performed this study to evaluate the safety and feasibility of transplantation with CRISPR/Cas9 CCR5 gene modified CD34+ hematopoietic stem/progenitor cells for patients that develop AIDS and hematological malignances. Patients will be treated with antiviral therapy (ART) to achieve undetectable HIV-1 virus in peripheral blood before conditioning. CD34+ cells from donors will be infused into the patients after treatment with CRISPR/Cas9 to ablate CCR5 gene.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the safety of the infusion of CD34+ cells which are treated with CRISPR/Cas9 to disrupt the CCR5 gene. The secondary objective is to evaluate the resistance to HIV-1(R5) in infected patients after infusion of modified CD34+ cells with or without an antiretroviral therapy interruption (ATI). After the transplantation, the reconstitution time and frequency of multi-lineage hematopoietic cell will be analyzed against previously reported HSCT in HIV-1 patients. After the detection of high CD4+ T cells reconstitution (over 600 cells/μL) and CCR5 negative cells (over 1%) in peripheral blood, subjects will undergo an ATI. HIV-1 RNA level and CD4+ cell counts will be monitored biweekly for at least one month.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 60, male of female;
2. Hematological neoplasms;
3. HIV-1 R5 tropic virus with no CXCR4-tropic or R5/X4 dual-tropic HIV;
4. On ART with undetectable HIV-1 level (<40gc/ml, HIV-1 RNA);
5. Availability of a consenting HLA-matched donor;
6. No cardiomyopathy or congestive heart failure;
7. CD4+ T-cell counts ≥200 cells/µL and ≤750 cells/µL;
8. Absence of psychosocial conditions and be willing to comply with study-mandated evaluations for 2 years;
9. Life expectancy of at least 1 year.

Exclusion Criteria:

1. Acute or chronic hepatitis B or hepatitis C infection;
2. Any cancer or malignancy other than hematological neoplasms;
3. Subject with CMV retinitis or other active CMV infection related diseases;
4. Subject with organ dysfunction;
5. Non-pregnant and non-nursing;
6. Drug or alcohol abuse or dependence;
7. Currently enrolled in another clinical trial or underwent cell therapy;
8. Donor incapable for HSPC mobilization;
9. in the opinion of the site investigator, would interfere with adherence to study requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2017-05-30 (Estimated); Primary Completion 2019-05-20 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
Persistence of CCR5 gene disruption in engrafted cells | 12 months
  Participants will be transplanted with CD34+ cells which are treated using the CRISPR/Cas9 system to disrupt CCR5 gene. The persistence of CCR5 gene disruption in engrafted cells will be evaluated by sequencing.

SECONDARY OUTCOMES:
CD34+ cell number | the first month
  The CD34+ cell number pre-infusion

OTHER OUTCOMES:
Gene disruption efficiency of bone marrow cells | Up to Month 12
  The percentage of disrupted CCR5 gene alleles in genome from bone marrow cells detected by sequencing.
CCR5 gene disruption efficiency of peripheral blood cells | Up to Month 12
  The percentage of disrupted CCR5 gene alleles in genome of peripheral blood cells by sequencing.
Hematopoietic cell engraftment | Up to Year 3
  Measurement of multi-lineage hematopoietic cell engraftment time after transplantation to evaluate the hematological recovery
HIV-1 RNA level | Up to Year 3
  Level change of HIV-1 RNA in plasma after transplantation
CD4+ T cell number | Up to Year 3
  Level change of the CD4+ T cell number after transplantation
The ratio change of CD4/CD8 | Up to Year 3
  The ratio change of CD4/CD8 in peripheral blood after transplantation
HIV-1 RNA levels during ATI | Every two weeks, until the end of ATI or up to 3 months
  HIV-1 RNA levels in plasma during ATI.
HIV-1 DNA level | Up to Month 12
  Changes of proviral DNA in PBMC pre- transplantation and 12 month post-transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- 307 Hospital of PLA (Affiliated Hospital of Academy to Military Medical Sciences), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu L, Wang J, Liu Y, Xie L, Su B, Mou D, Wang L, Liu T, Wang X, Zhang B, Zhao L, Hu L, Ning H, Zhang Y, Deng K, Liu L, Lu X, Zhang T, Xu J, Li C, Wu H, Deng H, Chen H. CRISPR-Edited Stem Cells in a Patient with HIV and Acute Lymphocytic Leukemia. N Engl J Med. 2019 Sep 26;381(13):1240-1247. doi: 10.1056/NEJMoa1817426. Epub 2019 Sep 11. PMID 31509667